CLINICAL TRIAL: NCT04450004
Title: A Randomized, Partially-Blinded, Dose-Ranging Phase 1 Study to Assess the Safety, Tolerability, and Immunogenicity of a Recombinant Coronavirus-Like Particle COVID 19 Vaccine in Adults 18-55 Years of Age
Brief Title: Safety, Tolerability and Immunogenicinity of a Coronavirus-Like Particle COVID-19 Vaccine in Adults Aged 18-55 Years.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medicago (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: CP-PRO-COVLP-019
Record Dates: First submitted 2020-06-18; First posted 2020-06-29 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: SARS-CoV 2

STUDY DESIGN:
Masking Description: Partially-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (9):
- Vaccine (3.75 µg) unadjuvanted (Experimental): • Group 1: 3.75 µg of the Coronavirus-Like Particle COVID-19 Vaccine
  Interventions: Biological: Intramuscular Vaccine
- Vaccine (3.75 µg) adjuvanted with CpG 1018 (Experimental): • Group 2: 3.75 µg of the Coronavirus-Like Particle COVID-19 Vaccine adjuvanted with CpG 1018
  Interventions: Biological: Intramuscular Vaccine
- Vaccine (3.75 µg) adjuvanted with AS03 (Experimental): • Group 3: 3.75 µg of the Coronavirus-Like Particle COVID-19 Vaccine adjuvanted with AS03
  Interventions: Biological: Intramuscular Vaccine
- Vaccine (7.5 µg) unadjuvanted (Experimental): • Group 4: 7.5 µg of the Coronavirus-Like Particle COVID-19 Vaccine unadjuvanted
  Interventions: Biological: Intramuscular Vaccine
- Vaccine (7.5 µg) adjuvanted with CpG 1018 (Experimental): • Group 5: 7.5 µg of the Coronavirus-Like Particle COVID-19 Vaccine adjuvanted with CpG 1018
  Interventions: Biological: Intramuscular Vaccine
- Vaccine (7.5 µg) adjuvanted with AS03 (Experimental): • Group 6: 7.5 µg of the Coronavirus-Like Particle COVID-19 Vaccine adjuvanted with AS03
  Interventions: Biological: Intramuscular Vaccine
- Vaccine (15 µg) unadjuvanted (Experimental): • Group 7: 15 µg of the Coronavirus-Like Particle COVID-19 Vaccine unadjuvanted
  Interventions: Biological: Intramuscular Vaccine
- Vaccine (15 µg) adjuvanted with CpG 1018 (Experimental): • Group 8: 15 µg of the Coronavirus-Like Particle COVID-19 Vaccine adjuvanted with CpG 1018
  Interventions: Biological: Intramuscular Vaccine
- Vaccine (15 µg) adjuvanted with AS03 (Experimental): • Group 9: 15 µg of the Coronavirus-Like Particle COVID-19 Vaccine adjuvanted with AS03
  Interventions: Biological: Intramuscular Vaccine

INTERVENTIONS:
Biological: Intramuscular Vaccine — Subjects will receive two intramuscular (IM) injections 21 days apart (Day 0 and Day 21), into the deltoid region of the alternating arm (each arm will be injected once), with their assigned vaccine.

SUMMARY:
The study will be a randomized, partially-blinded, prime-boost, staggered dose-escalation Phase 1 study intended to assess the safety, tolerability, and immunogenicity of the Coronavirus-Like Particle COVID-19 Vaccine at three dose levels (3.75 µg, 7.5 µg, and 15 µg VLP) unadjuvanted or adjuvanted with either CpG 1018 or AS03 in healthy adults 18 to 55 years of age, who have been tested for the absence of SARS-CoV-2 antibodies.

At each dose level, the vaccine will initially be administered to a small number of subjects. Vaccinations of the first 6 subjects at the lowest dose level will be staggered so that each vaccination must be performed at least 30 minutes apart. Vaccination of the remaining subjects at the same dose level and the next higher vaccine dose level will be administered with approval of the Independent Data Monitoring Committee (IDMC). The same process will be followed for the second vaccine administration. All subjects will be followed for a period of 12 months after the second administration of the vaccine for safety and immunogenicity testing at the end of the follow-up period.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria at the Screening (Visit 1) and/or Vaccination (Visit 2) visits to be eligible for participation in this study; no protocol waivers are allowed. All Investigator assessment-based judgements must be carefully and fully documented in the source documents:

1. Subjects must have read, understood, and signed the informed consent form (ICF) prior to participating in the study; subjects must also complete study-related procedures and communicate with the study staff at visits and by phone during the study;
2. At the Screening visit (Visit 1), male and female subjects must be 18 to 55 (has not yet had his/her 56th birthday) years of age, inclusive;
3. At Screening (Visit 1) and Vaccination (Visit 2), subject must have a body mass index (BMI) of ≥ 18.5 and < 25 kg/m2;
4. Subjects are considered by the Investigator to be reliable and likely to cooperate with the assessment procedures and be available for the duration of the study;
5. Subjects must be healthy (no clinically significant health concerns) as determined by medical history, physical examination, vital signs, and clinical laboratory tests. Investigator discretion will be permitted with this inclusion criterion;
6. Female subjects of childbearing potential must have a negative serum pregnancy test result at Screening (Visit 1) and a negative urine pregnancy test result at Vaccination (Visit 2 and Visit 4).

   Non-childbearing females are defined as:
   * Surgically-sterile (defined as bilateral tubal ligation, hysterectomy or bilateral oophorectomy performed more than one month prior to the first study vaccination); or
   * Post-menopausal (absence of menses for 12 consecutive months and age consistent with natural cessation of ovulation);
7. Female subjects of childbearing potential must use an effective method of contraception for one month prior to vaccination (Visit 2) and agree to continue employing highly effective birth control measures for at least one month after the last administration of the investigational product (or in the case of early termination, she must not plan to become pregnant for at least one month after her last study vaccination). The following relationship or methods of contraception are considered to be highly effective:

   * Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation:
   * Oral;
   * Intravaginal;
   * Transdermal;
   * Progestogen-only hormonal contraception associated with inhibition of ovulation:
   * Oral;
   * Injectable;
   * Implantable;
   * Intra-uterine device with or without hormonal release;
   * Vasectomised partner, provided that this partner is the sole sexual partner of the study participant and that the vasectomised partner has received a medical assessment of the surgical success;
   * Credible self-reported history of heterosexual vaginal intercourse abstinence prior to and for at least one month after the last administration of the investigational product ;
   * Female partner.

Exclusion Criteria:

Subjects who meet any of the following criteria at the Screening (Visit 1) and/or Vaccination (Visit 2) visits will not be eligible for participation in this study; no protocol waivers are allowed. All Investigator assessment-based judgements must be thoroughly documented in the source documents:

1. Clinically significant acute or chronic pulmonary (including but not limited to chronic obstructive pulmonary disease or asthma), cardiovascular (including but not limited to arterial hypertension, coronary artery disease, or congestive heart failure), renal, metabolic (including but not limited to type 2 diabetes), or other somatic (medical) or neuropsychiatric illness within 3 months prior to Screening (Visit 1), excessive alcohol use or drug abuse, as determined by medical history, physical examination, vital signs, and clinical laboratory tests.

   Investigator discretion is permitted with this exclusion criterion and must be carefully and fully documented in the source documents;
2. Any unexplained clinical syndrome (including, but not limited to, chronic fatigue syndrome, Raynaud's syndrome, unexplained pain syndromes such as fibromyalgia, etc.);
3. Acute disease defined as presence of any moderate or severe acute illness with or without a fever within 48 hours prior to Vaccination (Visit 2);
4. Prior exposure to SARS-CoV-2 as determined by detection of IgM or IgG antibodies against SARS-CoV-2 at Screening (Visit 1) and Vaccination (Visit 2);
5. Any confirmed or suspected current immunosuppressive condition or immunodeficiency, including cancer, human immunodeficiency virus (HIV), hepatitis B or C infection (subjects with a history of cured hepatitis B or C infection without any signs of immunodeficiency at present time are allowed). Investigator discretion is permitted with this exclusion criterion;
6. Current autoimmune disease (such as rheumatoid arthritis, systemic lupus erythematosus or multiple sclerosis). Investigator discretion is permitted with this exclusion criterion, and subjects may be eligible to participate with appropriate written justification in the source document (i.e. subjects with a history of autoimmune disease who are disease-free without treatment for three years or more, or on stable thyroid replacement therapy, mild psoriasis [i.e. a small number of minor plaques requiring no systemic treatment], etc.);
7. Administration of any medication or treatment that may alter the vaccine immune responses, such as:

   * Systemic glucocorticoids within one month prior to Vaccination (Visit 2). Inhaled, nasal, dermal, intraarticular, ophthalmic and other topical glucocorticoids are permitted;
   * Cytotoxic, antineoplastic, or immunosuppressant drugs - within 36 months prior to Vaccination (Visit 2);
   * Any immunoglobulin preparations or blood products, blood transfusion - within 6 months prior to Vaccination (Visit 2);
8. Administration of any vaccine within 30 days prior to Vaccination (Visit 2); planned administration of any vaccine during the study (up to blood sampling on Day 42 of the study). Immunization on an emergency basis during the study will be evaluated on case-by-case basis by the Investigator;
9. Administration of any other SARS-CoV-2 / COVID-19, or other experimental coronavirus vaccine at any time prior to or during the study;
10. Known current or previous laboratory-confirmed SARS-CoV-1 or SARS-CoV-2 / COVID 19 infection as documented by a positive PCR test or positive serological test;
11. Subjects at high risk of contracting SARS-CoV-2/COVID-19 infection, including but not limited to the individuals with known close contact of anyone with laboratory-confirmed SARS-CoV-2 / COVID-19 infection within 2 weeks prior to vaccine administration, those who traveled outside Canada for any duration within 30 days before the study vaccination, healthcare workers in acute care hospitals, rehabilitation hospitals, mental health hospitals, long term care facilities, emergency departments, and others who through their work must come into close face-to-face contact with their clients or patients (including, but not limited to, physiotherapists, dentists, hair dressers/barbers, etc.);
12. Use of any investigational or non-registered product within 30 days or 5 half-lives, whichever is longer, prior to Vaccination (Visit 2) or planned use during the study period;
13. Have a rash, dermatological condition, tattoos, muscle mass, or any other abnormalities at injection site that may interfere with injection site reaction rating. Investigator discretion will be permitted with this exclusion criterion;
14. Use of any prescription medication on a regular basis for more than 30 continuous days within the last 3 months, with the following exceptions:

    * Medications listed among the methods of contraception in inclusion criterion 7;
    * Subjects on stable thyroid replacement therapy, as noted in exclusion criterion 6.
15. Use of any prescription antiviral drugs with the intention of COVID-19 prophylaxis, including those that are thought to be effective for prevention of COVID-19 but have not been licensed for this indication, within one month prior to Vaccination (Visit 2);
16. Use of prophylactic medications (e.g. antihistamines [H1 receptor antagonists], nonsteroidal anti-inflammatory drugs [NSAIDs], systemic and topical glucocorticoids, non-opioid and opioid analgesics) within 24 hours prior to the Vaccination (Visit 2) to prevent or pre-empt symptoms due to vaccination;
17. History of allergy to any of the constituents of the Coronavirus-Like Particle COVID-19 Vaccine, vaccine adjuvants, or tobacco;
18. History of anaphylactic allergic reactions to plants or plant components (including fruits and nuts);
19. Currently smoke more than 10 cigarettes per month or any use of vaping products;
20. Subjects with a history of Guillain-Barré Syndrome;
21. Any female subject who has a positive or doubtful pregnancy test result prior to vaccination or who is lactating;
22. Subjects identified as an Investigator or employee of the Investigator or clinical site with direct involvement in the proposed study, or identified as an immediate family member (i.e. parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed study, or any employees of Medicago.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2020-07-10 (Actual); Primary Completion 2020-09-20 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Immediate adverse event (AEs) | 30 minutes
  Percentage, intensity, and relationship to vaccination of immediate adverse events (AEs)
Solicited local and systemic adverse events (AEs) | 7 days
  Percentage, intensity, and relationship to vaccination of solicited local and systemic adverse events (AEs) following each vaccination
Unsolicited adverse events (AEs) | 21 days
  Percentage, intensity, and relationship of unsolicited adverse events (AEs) following each vaccine administration
Serious adverse events (SAEs), adverse events (AEs) leading to withdrawal, adverse event of special interest (AESI) (including vaccine-enhanced disease) and deaths | 21 days
  Occurrences of serious adverse events (SAEs), adverse events (AEs) leading to withdrawal, adverse event of special interest (AESIs) (including vaccine-enhanced disease (VED)), and deaths following each vaccine administration
Safety labs | 3 days
  Number and percentage of subjects with normal and abnormal clinically significant urine, haematological and biochemical values prior to and 3 days following each vaccination.
Neutralizing antibody (Nab assay) response | 21 days
  Nab response induced by the vaccine against the SARS-CoV-2 virus
Specific Th1 cell-mediated immunity (CMI) response | 21 days
  Cell-mediated immunity (CMI) response induced by the vaccine against the SARS-CoV-2 virus after each vaccination, as measured by Interferon-gamma (IFN-γ) enzyme-linked immunospot (ELISpot)
Specific Th2 cell-mediated immunity (CMI) response | 21 days
  Cell-mediated immunity (CMI) response induced by the vaccine against the SARS-CoV-2 virus after each vaccination, as measured by Interleukin-4 (IL-4) ELISpot

SECONDARY OUTCOMES:
Serious adverse events (SAEs), adverse events (AEs) leading to withdrawal, adverse event of special interest (AESI) (including vaccine-enhanced disease) and deaths | Day 42 to 386
  Occurrences of serious adverse events (SAEs), adverse events (AEs) leading to withdrawal, adverse event of special interest (AESIs) (including vaccine-enhanced disease (VED)), and deaths from 22 days after the last vaccination up to the end of the study
Specific antibody response induced by the vaccine against the SARS-CoV-2 virus measured by total IgG and/or IgM levels | Day 21, 42, 201 and 386
  Specific antibody response induced by the vaccine against the SARS-CoV-2 virus, as measured by total IgG and/or IgM levels
Neutralizing antibody (Nab assay) response induced by the treatment groups against the SARS-CoV-2 virus | Day 201 and 386
  Neutralizing antibody (Nab assay) response induced by the treatment groups against the SARS-CoV-2 virus
Specific Th1 cell-mediated immunity (CMI) response induced by the vaccine against the SARS-CoV-2 virus | Day 201 and 386
  Specific Th1 cell-mediated immunity (CMI) response induced by the vaccine against the SARS-CoV-2 virus measured by IFN- γ ELISpot
Specific Th2 cell-mediated immunity (CMI) response induced by the vaccine against the SARS-CoV-2 virus | Days 201 and 386
  Specific Th2 cell-mediated immunity (CMI) response induced by the vaccine against the SARS-CoV-2 virus measured by IL-4 ELISpot.

OTHER OUTCOMES:
Specific cell-mediated immunity (CMI) response induced by the vaccine against the SARS-CoV-2 virus | Day 21, 201 and 386
  Specific cell-mediated immunity (CMI) response induced by the vaccine against the SARS-CoV-2 virus measured by the percentage of CD4+ T cells expressing functional markers
Specific antibody response induced by the vaccine against plant glycans | Day 21, 201 and 386
  Specific antibody response induced by the vaccine against plant glycans as measured by serum IgE levels directed against Cross-reactive Carbohydrate Determinants (CCD) MUXF3 using bromelain glycoprotein
Further characterization of the immune response and the safety profile of the Coronavirus-Like Particle COVID-19 Vaccine | Day 21, 42, 201, 386
  If deemed necessary, further characterization of the immune response and the safety profile of the Coronavirus-Like Particle COVID-19 Vaccine
Laboratory-confirmed SARS-CoV-2 infection | Day 0 to 386
  Occurrence(s) of laboratory-confirmed (virologic or serologic methods) SARS-CoV-2 infection (with or without symptoms
Characterization of the immune response of the Coronavirus-Like Particle COVID-19 Vaccine | Up to day 386
  • If deemed necessary, further characterization of the immune response of the Coronavirus-Like Particle COVID-19 Vaccine.

CONTACTS AND LOCATIONS:
Overall Officials: Brian J Ward, MD, Study Director — Medicago
Locations (2):
- Canada (2):
  - Syneos Health, Montreal, Quebec
  - Syneos Health, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ward BJ, Gobeil P, Seguin A, Atkins J, Boulay I, Charbonneau PY, Couture M, D'Aoust MA, Dhaliwall J, Finkle C, Hager K, Mahmood A, Makarkov A, Cheng MP, Pillet S, Schimke P, St-Martin S, Trepanier S, Landry N. Phase 1 randomized trial of a plant-derived virus-like particle vaccine for COVID-19. Nat Med. 2021 Jun;27(6):1071-1078. doi: 10.1038/s41591-021-01370-1. Epub 2021 May 18. PMID 34007070